CLINICAL TRIAL: NCT03325803
Title: Efficacy in Ablative Fractional Laser Assisted Photodynamic Therapy According to Ablative Depth for Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Song Ki-Hoon, Professor and chairman, Department of dermatology Dong-A University, College of medicine, Dong-A University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: DAUderma-08
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Actinic Dermatosis
Keywords: actinic keratosis; ablative fractional laser; photodynamic therapy; ablative depth; protoporphyrin IX
MeSH Terms: conditions — Keratosis, Actinic | interventions — Lidocaine; Prilocaine; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 150μm-AFL-PDT (Experimental)
  Interventions: Drug: lidocaine/prilocaine (5%) application; Device: 2940-nm Er:YAG AFL pretreatment; Drug: MAL application; Other: Measurements of the fluorescence intensity; Device: irradiation with red light-emitting diode lamp
- 350μm-AFL-PDT (Experimental)
  Interventions: Drug: lidocaine/prilocaine (5%) application; Device: 2940-nm Er:YAG AFL pretreatment; Drug: MAL application; Other: Measurements of the fluorescence intensity; Device: irradiation with red light-emitting diode lamp
- 500μm-AFL-PDT (Experimental)
  Interventions: Drug: lidocaine/prilocaine (5%) application; Device: 2940-nm Er:YAG AFL pretreatment; Drug: MAL application; Other: Measurements of the fluorescence intensity; Device: irradiation with red light-emitting diode lamp

INTERVENTIONS:
Drug: lidocaine/prilocaine (5%) application — For AFL pre-treatment, lidocaine/prilocaine (5%) cream (EMLA; Astra Pharmaceuticals, LP, Westborough, MA, USA) was applied to the treatment area under occlusion for 30 min
Device: 2940-nm Er:YAG AFL pretreatment — After the anaesthetic cream was removed, AFL therapy was performed using a 2940-nm Er:YAG AFL (Joule; Sciton Inc., Palo Alto, CA, USA) at 150 µm ablation depth, level 1 coagulation, 22% treatment density and a single pulse
Drug: MAL application — Immediately after AFL treatment, an approximately 1- mm-thick layer of MAL (Metvix, PhotoCure ASA, Oslo, Norway) was applied to the lesion and on 5 mm of surrounding normal tissue. Incubation time is 3 hours
Other: Measurements of the fluorescence intensity — After 3 hours of application with MAL, saline wash was performed and fluorescence imaging analysis was performed with ultraviolet examination light (model 31602,356 nm; Burton Medical Products Crop.) at 10 cm height above the base of each lesion. The red fluorescence (610 nm-700 nm) was separated and extracted by Matlab program and then used to measure the amount of 633 nm fluorescence of protoporphyrin IX.
Device: irradiation with red light-emitting diode lamp — After incubation for 3 hours, the dressing and cream were removed, and the area was cleansed with saline. The area was irradiated with a red light-emitting diode lamp (Aktilite CL 128; PhotoCure ASA, Oslo, Norway) with peak emission at 632 nm, placed 5 cm away from the skin surface, and a total light dose of 37 J/cm-2. All patients wore protective goggles during illumination.

SUMMARY:
Er:YAG ablative fractional laser-assisted photodynamic therapy (AFL-PDT) has shown significant benefit for the treatment of actinic keratosis(AK). Er:YAG ablative fractional laser ablates the epidermis and dermis without significant thermal injury, creating microscopic ablation zones (MAZ) in the portion of the skin that the laser is applied to. The formed MAZ depends on the laser parameters such as laser depth, laser density and laser passes, which affect the treatment outcome.

DETAILED DESCRIPTION:
The investigators aimed to investigate whether the use of increased laser ablative depth affects the efficacy, side effects, cosmetic outcomes, and PPIX accumulation of AFL-PDT for facial AK in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Korean patients aged ≥ 18 years who had biopsy-confirmed Actinic keratosis lesions

Exclusion Criteria:

* photosensitivity disorder patients
* lactating or pregnant women
* patients with porphyria or a known allergy to any of the constituents of the MAL cream and lidocaine
* patients with systemic disease, history of malignant melanoma, tendency of melasma development or keloid formation, any AK treatment of the area in the previous 4 weeks, or any conditions associated with a risk of poor protocol compliance; and patients on immunosuppressive treatment

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Differences of short-term complete response rates between 3 groups | Short-term complete response rates were evaluated at 3 months after treatment
  Lesion responses were classified as either a complete response (complete disappearance of the lesion) or a noncomplete response (incomplete disappearance)
Differences of long-term complete response rates between 3 groups | Long-term complete response rates were evaluated at 12 months
  In all cases of complete response, the patients were reviewed at 12 months to check for recurrence. Recurrence was assessed by inspection, dermoscopy, photography, palpation, and histologic findings. For the histopathologic evaluation of treatment response, at the 12-month follow-up visit, a 3-mm punch biopsy of the treated AK lesion was performed in all cases of clinically incomplete response.
Difference of the recurrence rates between 3 groups | Recurrence rates were evaluated respectively at 12 months after treatment
  In all cases of complete response, the patients were reviewed at 12 months to check for recurrence. Recurrence was assessed by inspection, dermoscopy, photography, palpation, and histologic findings. For the histopathologic evaluation of treatment response, at the 12-month follow-up visit, a 3-mm punch biopsy of the treated AK lesion was performed in all cases of clinically incomplete response.
Differences of the fluorescence intensity between 3 groups | After 3 hours of application with MAL, fluorescence intensity imaging was assessed 10 minutes before illumination.
  After 3 hours of application with MAL, Fluorescence imaging analysis was performed on treatment area with ultraviolet examination light (model 31602,356 nm; Burton Medical Products Crop.) at 10 cm height above the base of each lesion. The red fluorescence was separated and extracted by Matlab program and then used to measure the amount of 633 nm fluorescence of protoporphyrin IX.

SECONDARY OUTCOMES:
Differences of cosmetic outcomes between 3 groups | The overall cosmetic outcome was assessed 12 months after treatment
  Cosmetic outcomes were graded as excellent (slight redness or pigmentation change), good (moderate redness or pigmentation change), fair (slight-to-moderate scarring, atrophy, or induration), or poor (extensive scarring, atrophy, or induration)
Difference of adverse events (erythema, post-inflammatory hyperpigmentation, edema, itching, oozing, bleeding) rates between 3 groups | Within 12 months after each treatment
  Adverse events reported by the patient were noted at each follow-up visit, including severity, duration and need for additional therapy. All events due to PDT were described as phototoxic reactions (i.e., erythema, post-inflammatory hyperpigmentation, oedema, itching, oozing, bleeding and so forth).

CONTACTS AND LOCATIONS:
Locations (1):
- Dong-A University, Busan, Seo-gu, Korea, Republic Of, 602-715, South Korea

IPD SHARING:
Plan to Share IPD: No